CLINICAL TRIAL: NCT04063514
Title: The Use of Focused Ultrasound and DCE K-trans Imaging to Evaluate Permeability of the Blood-Brain Barrier
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICSS-2018-001
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Low Grade Glioma of Brain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Focused Ultrasound (Experimental): The ultrasound treatment will last either 1 hour or 20 minutes total time for the DWL device or Brainsonix Focused Ultrasound Device, respectively.
  Interventions: Other: Focused Ultrasound

INTERVENTIONS:
Other: Focused Ultrasound — With focused ultrasound, there is an expected accentuation of local perfusion and potential temporary opening of the blood brain barrier with the aim is to provide better delivery of therapeutic agents including medication, particulates and cellular elements for treatment of neoplastic, inflammatory and degenerative brain diseases. The present study seeks to investigate differences in perfusion between areas treated and untreated by this modality in order to further explore its use in clinical application for the treatment of brain disease.

SUMMARY:
The limitation of treating intrinsic brain pathologies has been circumvented with neurosurgical techniques; however, less invasive approaches may be desirable particularly for widespread or multifocal disease and when long term and repetitive administration is required. This study seeks to investigate the efficacy of focused ultrasound.

Patients with either low grade gliomas or neurodegenerative dementias will be evaluated for study candidacy.

There are no immediate benefits for patients who choose to participate; however, the information gained from this study will contribute to the research base and help patients in similar situations in the future.

DETAILED DESCRIPTION:
Treatment of intrinsic brain diseases is challenging because brain barrier (BBB) limits the delivery of drugs, particulates and cellular elements such as stem cells to the central nervous system (CNS). This limitation is often circumvented with neurosurgical techniques, however, less invasive approaches may be desirable particularly for widespread or multifocal disease and when long term and repetitive administration is required.

The diagnosis for the participants will be either low grade gliomas. A baseline fMRI and follow up routine fMRI's will be taken and evaluated for any changes in perfusion. During the scans, The ultrasound placement will last for one hour.

This study seeks to investigate the efficacy of focused ultrasound in opening the blood brain barrier. This physiological effect would have significant clinical applications. The ability to open the blood brain barrier has the potential to revolutionize the delivery of therapeutic agents to the brain, allowing for more localized and efficient delivery. There are no immediate benefits for patients who choose to participate; however, the information gained from this study will contribute to the research base and help patients in similar situations in the future.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing routine, repetitive MRI scanning for monitoring low grade gliomas
* 18 or older

Exclusion Criteria:

• Cognitive decline with mild cognitive impairment (Clinical Dementia Rating stage 0.5) through moderate dementia CDR stages 1 and 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE) & Serious Adverse Event (SAE) Reporting | 24 hours
  Per protocol, any suspected adverse events possibly related to the study protocol (e.g., itching, dizziness, headache, or neurological problems) will be tracked and monitored. In the event of a high-grade or serious adverse event, such event will be reported immediately and the study will be discontinued.
functional Magnetic Resonance Imaging (fMRI) | 3 hours
  Some functional neuroimaging scans (e.g., high resolution T1-weighted images; Arterial Spin Labeling [ASL]; Dynamic Contrast Enhanced [DCE] perfusion sequences; post-contrast T1-weighted images, Susceptibility Weighted Imaging [SWI], T2 weighted imaging, and T2 Flair) will be used to evaluate longitudinal changes in perfusion as an efficacy measure. The scans will be acquired within one hour before and after the study procedures of focused transcranial ultrasound and infusion of definity microbubbles. Voxel-based comparisons showing perfusion values relative to the acquired data range will be used for quantification and comparison of baseline and post-procedure scans.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, M.D., Principal Investigator — Neurologist, NAOWLA
Locations (1):
- Neurological Associates of West LA, Santa Monica, California, United States

REFERENCES:
- [Background] McDannold N, Vykhodtseva N, Hynynen K. Targeted disruption of the blood-brain barrier with focused ultrasound: association with cavitation activity. Phys Med Biol. 2006 Feb 21;51(4):793-807. doi: 10.1088/0031-9155/51/4/003. Epub 2006 Jan 25. PMID 16467579
- [Background] McDannold N, Vykhodtseva N, Hynynen K. Use of ultrasound pulses combined with Definity for targeted blood-brain barrier disruption: a feasibility study. Ultrasound Med Biol. 2007 Apr;33(4):584-90. doi: 10.1016/j.ultrasmedbio.2006.10.004. PMID 17337109
- [Background] Hynynen K, McDannold N, Vykhodtseva N, Jolesz FA. Noninvasive MR imaging-guided focal opening of the blood-brain barrier in rabbits. Radiology. 2001 Sep;220(3):640-6. doi: 10.1148/radiol.2202001804. PMID 11526261
- [Background] Hynynen K, McDannold N, Sheikov NA, Jolesz FA, Vykhodtseva N. Local and reversible blood-brain barrier disruption by noninvasive focused ultrasound at frequencies suitable for trans-skull sonications. Neuroimage. 2005 Jan 1;24(1):12-20. doi: 10.1016/j.neuroimage.2004.06.046. PMID 15588592
- [Background] Hynynen K, McDannold N, Vykhodtseva N, Raymond S, Weissleder R, Jolesz FA, Sheikov N. Focal disruption of the blood-brain barrier due to 260-kHz ultrasound bursts: a method for molecular imaging and targeted drug delivery. J Neurosurg. 2006 Sep;105(3):445-54. doi: 10.3171/jns.2006.105.3.445. PMID 16961141
- [Background] Treat LH, McDannold N, Vykhodtseva N, Zhang Y, Tam K, Hynynen K. Targeted delivery of doxorubicin to the rat brain at therapeutic levels using MRI-guided focused ultrasound. Int J Cancer. 2007 Aug 15;121(4):901-7. doi: 10.1002/ijc.22732. PMID 17437269
- [Background] Schlachetzki F, Holscher T, Koch HJ, Draganski B, May A, Schuierer G, Bogdahn U. Observation on the integrity of the blood-brain barrier after microbubble destruction by diagnostic transcranial color-coded sonography. J Ultrasound Med. 2002 Apr;21(4):419-29. doi: 10.7863/jum.2002.21.4.419. PMID 11934099
- [Background] Yoshikawa K, Davies A. Safety of ProHance in special populations. Eur Radiol. 1997;7 Suppl 5:246-50. doi: 10.1007/pl00006901. PMID 9370552
- [Background] Semelka RC, Ramalho J, Vakharia A, AlObaidy M, Burke LM, Jay M, Ramalho M. Gadolinium deposition disease: Initial description of a disease that has been around for a while. Magn Reson Imaging. 2016 Dec;34(10):1383-1390. doi: 10.1016/j.mri.2016.07.016. Epub 2016 Aug 13. PMID 27530966
- [Background] Todd DJ, Kay J. Gadolinium-Induced Fibrosis. Annu Rev Med. 2016;67:273-91. doi: 10.1146/annurev-med-063014-124936. PMID 26768242
- [Result] McDannold N, Vykhodtseva N, Raymond S, Jolesz FA, Hynynen K. MRI-guided targeted blood-brain barrier disruption with focused ultrasound: histological findings in rabbits. Ultrasound Med Biol. 2005 Nov;31(11):1527-37. doi: 10.1016/j.ultrasmedbio.2005.07.010. PMID 16286030

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04063514/Prot_ICF_000.pdf